CLINICAL TRIAL: NCT03088618
Title: A Multi-center, Non-randomized, Open, Single-arm Confirmatory Clinical Study to Evaluate the Safety and Efficacy of Surgical Material for Nasal Septoplasty in Septal Deformity Patients With Nasal Obstruction
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of Surgical Material for Nasal Septoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: T&R Biofab Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNRBIOFAB-CTS01
Record Dates: First submitted 2017-02-09; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Septal Deformity; Nasal Obstruction
Keywords: Nasal obstruction; Septal deformity; Septoplasty; TnR Mesh; polycaprolactone
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with septal deformity (Experimental): To evaluate the safety and efficacy of surgical material for nasal septoplasty in septal deformity patients with nasal obstruction
  Interventions: Procedure: Nasal septoplasty

INTERVENTIONS:
Procedure: Nasal septoplasty — Type of surgery

SUMMARY:
The purpose of this clinical trial is to evaluate safety and efficacy of TnR mesh for patients who need nasal septoplasty for septal deformity with nasal obstruction.

DETAILED DESCRIPTION:
Nasal obstruction is a nasal disease commonly seen in the area of otolaryngology, and major symptoms include nasal congestion, rhinitis, and etc.

Nasal septoplasty is a surgery performed to improve above symptoms of nasal obstruction and so far, many surgical technique have been studied. All surgical techniques aimed to improve breathing through the nasal cavity by supporting the end of nose using surgical materials such as autologous bone or nonabsorbable material.

In the case of autologous bone transplantation, safety is ensured, but there is a limitation since it causes deficiency of the donor site, and the nasal septum may be altered by a modification of the implanted tissue.

In the case of nonabsorbable materials, there is a high risk of side effects such as hyposmia, septal perforation, and occurrence of boil.

TnR mesh, as a surgical material for nasal septoplasty has a sufficient flexural strength to support the nasal septum and to overcome the force of returning to a deviated state prior to surgery.

Animal tests have shown that TnR mesh well supports the nasal septum after surgery and the surrounding tissue is well fused between the pores without inflammatory responses. Based on above results, a clinical trial was planned to evaluate the efficacy and safety of TnR mesh as a material for nasal septoplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with nasal septal deformity who require surgical treatment
2. Females of childbearing potential must have a negative urine pregnancy test, and must not plan to become pregnant during the course of the study.

Exclusion Criteria:

1. Known allergic reaction to medical devices(TnR mesh) of the clinical trial
2. Pregnancy or lactation

   - Before screening
3. History of surgery in nasal or paranasal sinuses before screening
4. History of radiation treatment at Head and neck
5. History of having participated in other clinical trial of a drug/ a medical device within three months

   - Screening point
6. Patients with untreated nasal bone fraction or trauma of nasal
7. Patients with surgical site infection caused by nasal bone fraction or trauma
8. Patients with untreated a perforation of septum, a sinusitis, a nasal cavity polyposis, a nasal cavity sarcoidosis, nasal valve collapse or wegener's granulomatosis
9. Patients with inflammation in a nasal cavity
10. Patients with sarcoma or carcinoma in a nasal cavity
11. Patients with asthma
12. Patients with untreated palate-facial disfigurements or cleft palate
13. Patients with systemic inflammatory disease
14. Patients with sepsis

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
NOSE total scores at 12 weeks after the surgery | 12 weeks
  The change in NOSE total scores of the 12th week after the surgery

SECONDARY OUTCOMES:
NOSE total scores | 4 weeks
  The change in NOSE total scores 4 weeks after the surgery
NOSE score by topic | 4 and 12 weeks
  NOSE score by topic 4, 12 weeks after the surgery
Acoustic rhinometry results(cross-sectional sum) | 4 and 12 weeks
  Changes in bilateral nasal cavity cross sectional sum in acoustic rhinometry results 4, 12 weeks after the surgery
Acoustic rhinometry results(volume sum) | 4 and 12 weeks
  Changes in bilateral nasal cavity volume sum in acoustic rhinometry results 4, 12 weeks after the surgery
CT images(cross sectional area) | 12 weeks
  Changes in nasal cavity cross-sectional area in CT images 12 weeks after the surgery
CT images(ratio of convex to concave side) | 12 weeks
  Changes in nasal cavity raio of convex to concave side of cross-sectional area in CT images 12 weeks after the surgery
CT images(nasal septum angle) | 12 weeks
  Changes in nasal septum angle in CT images 12 weeks after the surgery
Ratio of improvement regarding symptoms | 12 weeks
  Ratio of improvement regarding symptoms 12 weeks after surgery
Level of satisfaction of patients | 12 weeks
  Satisfaction score(used visual analogue scale) of subject 12 weeks after surgery

OTHER OUTCOMES:
Deviant-cases | 12 weeks
  A follow-up will be performed after the surgery until the end of the clinical trial period. Any newly occurred or worsen symptoms will be recorded.
  Preparation content: Deviant-cases name, expression date, disappearance date, severity, gravity, results, a relationship between a medical device, a treatment, a status(remove or not).
  All deviant-cases are standardized as System Organ Class (SOC) and Preferred Term (PT) according to Medical Dictionary for regulatory activities (MedDRA). The analysis of deviant-case is based on the Treatment Emergent Adverse Event (TEAE). The percentage and the number of deviant cases and abnormal reactions to the device will be proposed as well as the 95 % of confidence interval of the incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Sung-won Kim, professor, Study Director — The Catholic University of Korea; Se-Hwan Hwang, professor, Study Director — The Catholic University of Korea Bucheon St.Mary's Hospital
Locations (2):
- South Korea (2):
  - The Catholic University of Korea, Bucheon-si, Gyeonggi-do
  - The Catholic University of Korea, Seoul ST. Mary's hospital, Seoul, Seocho-gu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Surowitz J, Lee MK, Most SP. Anterior Septal Reconstruction for Treatment of Severe Caudal Septal Deviation: Clinical Severity and Outcomes. Otolaryngol Head Neck Surg. 2015 Jul;153(1):27-33. doi: 10.1177/0194599815582176. Epub 2015 Apr 16. PMID 25883105
- [Background] Kim JH, Kim DY, Jang YJ. Outcomes after endonasal septoplasty using caudal septal batten grafting. Am J Rhinol Allergy. 2011 Jul-Aug;25(4):e166-70. doi: 10.2500/ajra.2011.25.3648. PMID 21819753
- [Background] Rimmer J, Ferguson LM, Saleh HA. Versatile applications of the polydioxanone plate in rhinoplasty and septal surgery. Arch Facial Plast Surg. 2012 Sep-Oct;14(5):323-30. doi: 10.1001/archfacial.2012.147. PMID 22986938
- [Background] Boenisch M, Nolst Trenite GJ. Reconstruction of the nasal septum using polydioxanone plate. Arch Facial Plast Surg. 2010 Jan-Feb;12(1):4-10. doi: 10.1001/archfacial.2009.103. PMID 20083734
- [Background] Kahveci OK, Miman MC, Yucel A, Yucedag F, Okur E, Altuntas A. The efficiency of Nose Obstruction Symptom Evaluation (NOSE) scale on patients with nasal septal deviation. Auris Nasus Larynx. 2012 Jun;39(3):275-9. doi: 10.1016/j.anl.2011.08.006. Epub 2011 Aug 31. PMID 21885221
- [Background] Stewart MG, Smith TL, Weaver EM, Witsell DL, Yueh B, Hannley MT, Johnson JT. Outcomes after nasal septoplasty: results from the Nasal Obstruction Septoplasty Effectiveness (NOSE) study. Otolaryngol Head Neck Surg. 2004 Mar;130(3):283-90. doi: 10.1016/j.otohns.2003.12.004. PMID 15054368
- [Background] Kim JN, Choi HG, Kim SH, Park HJ, Shin DH, Jo DI, Kim CK, Uhm KI. The efficacy of bioabsorbable mesh as an internal splint in primary septoplasty. Arch Plast Surg. 2012 Sep;39(5):561-4. doi: 10.5999/aps.2012.39.5.561. Epub 2012 Sep 12. PMID 23094256
- [Background] Garcia LB, Oliveira PW, Vidigal Tde A, Suguri Vde M, Santos Rde P, Gregorio LC. Caudal septoplasty: efficacy of a surgical technique-preliminary report. Braz J Otorhinolaryngol. 2011 Mar-Apr;77(2):178-84. doi: 10.1590/s1808-86942011000200007. PMID 21537619
- [Background] Erickson B, Hurowitz R, Jeffery C, Ansari K, El Hakim H, Wright ED, Seikaly H, Greig SR, Cote DW. Acoustic rhinometry and video endoscopic scoring to evaluate postoperative outcomes in endonasal spreader graft surgery with septoplasty and turbinoplasty for nasal valve collapse. J Otolaryngol Head Neck Surg. 2016 Jan 12;45:2. doi: 10.1186/s40463-016-0115-9. PMID 26754620
- See also: SIDS Initial Assessment Report — http://webnet.oecd.org/hpv/UI/handler.axd?id=2ccdc186-93a9-47cd-b91d-26789738233d